CLINICAL TRIAL: NCT02910349
Title: Novel Cardiac Imaging Prognostic Markers of Clinical Outcome in Patients With Chronic Aortic Regurgitation - Echocardiography and Magnetic Resonance
Brief Title: Novel Cardiac Imaging Prognostic Markers of Clinical Outcome in Patients With Chronic Aortic Regurgitation
Acronym: MOLLI-GLS-Hx
Status: Completed | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government); General University Hospital, Prague (Other); VZW Cardiovascular Research Center Aalst (Other); University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Radka Kockova, Dr Radka Kockova MD, PhD, Institute for Clinical and Experimental Medicine
Other Study IDs: 00023001
Record Dates: First submitted 2016-02-22; First posted 2016-09-22 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Aortic Valve Disorder
Keywords: valvular hear disease; echocardiography; magnetic resonance; global longitudinal strain; T1 relaxation time
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Myocardial biopsy specimen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Severe aortic regurgitation is a common valvular heart disease with prevalence of approximately 1%, affecting rather younger patients. The surgical treatment is the only causal treatment; it is recommended in patients with severe symptomatic aortic regurgitation. The optimal timing of the surgery is crucial because there is a certain risk of perioperative mortality and most patients require lifelong anticoagulation therapy. It is widely accepted, that asymptomatic patients with severely dilated left ventricle with systolic impairment have worse postoperative prognosis. We aim to evaluate native myocardial T1 relaxation time derived from cardiac magnetic resonance and global longitudinal left ventricular strain measured by echocardiography. These parameters are related to diffuse myocardial fibrosis and we expect to identify the cut off values, which correlate with further clinical course. This might enable better timing of the surgical treatment with the optimal postoperative left ventricular reverse remodelling and improved patient prognosis.

DETAILED DESCRIPTION:
Introduction:

Chronic aortic regurgitation is a common valvular heart disease with prevalence of approximately 1% in European population; affecting rather younger patients. The most common causes of chronic aortic regurgitation in developed countries are calcific aortic valve disease and bicuspid aortic valve. Another relatively frequent cause of the chronic aortic regurgitation is the aortic root dilation, which is genetically determined and it is also frequently diagnosed in younger patients. According to current guidelines for valvular heart disease, surgical treatment is recommended for patients with the severe symptomatic aortic regurgitation and for patients with the severe asymptomatic aortic regurgitation when left ventricular ejection fraction (LV EF) is < 50% or if other cardiothoracic surgery is planned (Class I). Current guidelines also recommend considering surgical strategy (Class IIa) in asymptomatic patients with severe aortic regurgitation, left ventricular ejection fraction (LV EF) ≥ 50% and left ventricular end-systolic diameter > 50 mm or indexed diameter > 25 mm/m2. There are two reasons for considering this earlier surgical treatment. Surgical techniques and perioperative treatment have improved recently and postoperative patient outcome are significantly better. There is also strong evidence that left ventricular (LV) diameter decreases shortly after surgery but left ventricular ejection fraction (LV EF) remains unchanged in majority of patients and left ventricular ejection fraction (LV EF) is one of the main determinants of patient's future quality of life and life expectancy. However, surgical correction might be indicated too late in clinical practice, typically in women. The Mayo Clinic authors group reported that women exhibit an excess late mortality compared to male population. They showed that women were severely symptomatic at the time of surgery compare to male population where left ventricular (LV) enlargement was more frequent. Bonow at al reported 33% incidence of clinical events, death and deterioration of left ventricular ejection fraction (LV EF), in natural history of asymptomatic patients with severe aortic regurgitation and preserved left ventricular ejection fraction (LV EF).

The optimal timing of surgical treatment is crucial but it has not been clearly established yet. New methods of identifying subclinical left ventricular (LV) function impairment are needed for better timing of the surgical strategy. Clinical follow-up with routine echocardiography study is recommended every 6 to12 months in patients with severe asymptomatic aortic regurgitation because sudden deterioration of left ventricular (LV) function might occur and we aim to operate on our patients before this happens. It is clear other parameters are needed than only left ventricular ejection fraction (LV EF) and left ventricular (LV) size. Diffuse myocardial fibrosis is a common feature of pathophysiology of the chronic left ventricular (LV) overload. Left ventricular ejection fraction (LV EF) and left ventricular (LV) size are less sensitive and non-specific markers of this process. Fortunately several novel methods of non-invasive quantification of the diffuse myocardial fibrosis have been introduced recently. The most promising method is the magnetic resonance imaging (MRI) - derived T1 relaxation time mapping introduced by Messroghli in 2004, Modified Look-Locker inversion recovery (MOLLI) sequence. Based on published data, MRI derived native T1 relaxation time is a reliable marker of diffuse myocardial fibrosis. The native T1 relaxation time with cut off value of ≥ 1010 ms is an accurate marker of extensive (>30%) myocardial fibrosis with high sensitivity and specificity (Ss=90%, Sp=73%, area under curve (AUC) =0.82). Extracellular myocardial volume (ECV) calculated from MOLLI sequence is also a sensitive marker of diffuse myocardial fibrosis and extracellular myocardial volume (ECV) cutoff value of ≥ 0.315 showed high accuracy to identify extensive (> 30%) myocardial collagen content (Ss=80%, Sp=90%, AUC =0.85). Speckle tracking echocardiography is another promising imaging method for diffuse myocardial fibrosis. Two-dimensional LV global longitudinal strain (GLS) has a potential to discover subclinical left ventricular (LV) functional impairment

Project Plan:

1. All patients will be scanned by MRI including Modified Look-Locker inversion recovery (MOLLI) within one week after inclusion and all complete and anonymized studies will be sent to CoreLab in IKEM. Off-line analysis will consist of the left and right ventricle volumetric and ejection fraction assessment. The aortic regurgitation will be measured using methods of flow sequence at sinotubular junction level (phantom correction required) and ventricular stroke volume difference. Modified Look-Locker inversion recovery (MOLLI) sequence will be acquired before, 10 and 15 minutes after contrast agent administration. T1 relaxation time will be measured within interventricular septum and ECV will be calculated from T1 relaxation time of the myocardium and the blood pool. Off-line analysis will be performed by two independent operators blinded to clinical and ECHO findings and intra- and inter-observer variability will be calculated.
2. All patients will undergo 2-D and 3-D transthoracic echocardiography within one week after inclusion and every six months during follow-up in each participating centre. All full volume anonymized studies will be sent to the CoreLab in IKEM. Off-line analysis of the left ventricular ejection fraction (LV EF),left ventricular (LV) volume, left ventricular (LV) mass, speckle tracking left ventricular (LV) global longitudinal strain (GLS), radial strain and left ventricular (LV) twist will be performed by two independent operators in a blinded fashion. Similarly aortic regurgitation grade will be assessed by two operators using colour Doppler, vena contracta measurement, and Doppler flow measurements. Inter- and intra-observer variability will be than calculated.
3. In all patients 12-lead electrocardiogram (ECG) will be recorded and blood sample will be taken during each visit. Brain natriuretic peptide serum level will be measured routinely at each participating centre. One blood sample will be stored frozen at -80 C° for further analysis including for example galectin levels, etc. This specific analysis will be performed in 1.Faculty of Medicine Charles University in Prague under the supervision of Prof. Sedmera.
4. Sub-study.

   1. All patients who will be scheduled for aortic valve surgery during follow-up (strictly according to current guidelines) will undergo perioperative myocardial needle biopsy from interventricular septum in each participating centre. All myocardial samples will be processed and analysed in 1.Faculty of Medicine Charles University in Prague under the supervision of Prof. Sedmera.
   2. All patients who will be scheduled for aortic valve surgery during follow-up will undergo repeat magnetic resonance imaging (MRI) study including Modified Look-Locker inversion recovery (MOLLI) sequence within 1-3 months prior to the operation and 6-12 month after the operation. The complete study will be repeated as described above. Postoperative left ventricular (LV) remodelling will be precisely assessed by off-line analysis. A correlation of the left ventricular (LV) remodelling and preoperative regurgitation grade as assessed by magnetic resonance imaging (MRI) and echocardiography (ECHO) will be calculated. Postoperative left ventricular (LV) remodelling will be also correlated with preoperative T1 myocardial relaxation time, extracellular volume (ECV) and global longitudinal strain (GLS).

Project Hypothesis:

1. We hypothesize that the increased native T1 longitudinal relaxation time as assessed by T1 mapping (Modified Look-Locker inversion recovery sequence) > 1010 ms and decreased global longitudinal strain (GLS) < 17 % are novel potent prognostic markers of clinical deterioration in patients with moderate to severe and severe chronic asymptomatic aortic regurgitation despite preserved left ventricular ejection fraction (LV EF).
2. We hypothesize that inter- and intra-observer variability of the aortic regurgitation severity assessment will be lower for the magnetic resonance imaging (MRI) study than for the echocardiography (ECHO) study.
3. We hypothesize that the degree of postoperative left ventricular (LV) recovery (decrease of the left ventricular (LV) volume and left ventricular (LV) mass) will correlate better with preoperative magnetic resonance imaging (MRI) regurgitation grade assessment rather than with echocardiography (ECHO) derived grade.

CoreLab The CoreLab will be located in Institute for Clinical and Experimental Medicine (IKEM) centre. All full volume anonymized magnetic resonance imaging (MRI) and 2-D and 3-D echocardiography (ECHO) studies will be sent to this CoreLab for off-line analysis. Two independent operators, specialists in the field of magnetic resonance imaging (MRI) and echocardiography (ECHO), will review all studies in a fully blinded fashion. One operator will repeat the analysis at least one month after the first reading. Inter- and intra-individual variability will then be calculated.

Myocardial biopsy and histology Myocardial sample will be obtained by experienced surgeon in all patients undergoing cardiothoracic surgery of the aortic valve. Under visual control a deep myocardial needle (SuperCore™ Semi-Automatic Biopsy Instrument 16 gauge x 9 cm) biopsy will be performed from the basal interventricular septum via the left ventricular outflow tract approach. A myocardial sample will be immersed immediately in 10% buffered formalin, embedded in paraffin blocks and later on sectioned at 3 micrometres (μm) thickness and stained with Picrosirius Red (PSR). PSR is a collagen specific stain and is an optimal tool for collagen quantification using normal light and also polarized light, which is helpful to distinguish between new and more matured collagen fibres. Percentage of myocardial fibrosis will be calculated as the ratio of Picrosirius Red (PSR)-positive area over total area using Image J software with differential thresholding. Histology analysis will be performed by experienced specialist on this field in a fully blinded fashion.

Laboratory analysis Fasting blood samples will be obtained during each visit and serum level of Hemoglobin, C-reactive protein, Hemoglobin A1c, Creatinine and Glucose level, Brain Natriuretic Peptide, Galectin 1 and 3 level will be measured. Creatinine clearance will be calculated using Cockcroft-Gault equation. One sample of frozen plasma will be stored for further analysis (but not for genetic analysis).

Number of included patients 100 - 150 patients in total.

Data Collection Patient data will be collected in one database system shared on-line with all centres. It will require an identification code for a patient and a centre. Under no circumstances will the patient data such as name, identification number (ID), address or other contact details be collected.

Study duration 2016 - 2022 (2 years recruitment + 5 years follow-up)

ELIGIBILITY:
Inclusion Criteria

1. Chronic asymptomatic aortic regurgitation grade 3 (moderate to severe) and grade 4 (severe)
2. No indication for the surgical treatment at the time of enrolment
3. LV EF ≥ 50 %
4. Absence of more than mild concomitant valve disease or complex congenital heart disease

Exclusion Criteria

1. Age < 18 years
2. Clearance Creatinine < 30 mL/min
3. Contraindication of magnetic resonance (implanted active device, ferromagnetic implant incompatible with magnetic resonance scanner, aneurysm clip, metallic fragment in the eye or near sensitive tissue)
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with grade 3 to 4 aortic regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Indication for aortic regurgitation surgical correction | within 7 years of follow-up
  number of participants undergoing valve surgery
Echocardiography (ECHO) - left ventricular (LV) end-systolic diameter (ESD) > 50 mm | each visit (6 months) within 7 years
  all participants
Echocardiography (ECHO) - left ventricular ejection fraction (LV EF) < 50 % finding | each visit (6 months) within 7 years
  all participants
Clinical symptoms occurrence such as dyspnoea class I (New York Heart Association (NYHA) | within 7 years of follow-up
  all participants
Arrhythmia (non-sustained or sustained ventricular tachycardia, ventricular ectopic beats > 10%, atrial fibrillation) | within 7 years of follow-up
  all participants
Hospitalization for heart failure symptoms | within 7 years of follow-up
  all participants
Laboratory findings: Brain natriuretic peptide (BNP) elevation > 150 ng/L | within 7 years of follow-up
  all participants
Cardiovascular death | within 7 years of follow-up
  all participants
Cumulative endpoint of all the above | within 7 years of follow-up
  all participants

SECONDARY OUTCOMES:
Echocardiography (ECHO) - Increase of left ventricular (LV) end-systolic diameter of > 10 mm in an individual patient without surgery | within 7 years
  in unoperated participants
Echocardiography (ECHO) - Increase of left ventricular (LV) end-diastolic diameter of > 15 mm in an individual patient without surgery | within 7 years
  in unoperated participants
Echocardiography (ECHO) - Decrease of global longitudinal strain (GLS) of > 5 % in an individual patient without surgery | within 7 years
  in unoperated participants
Echocardiography (ECHO) - Increase of left ventricular (LV) mass index of > 10 % in an individual patient without surgery | within 7 years
  in unoperated participants
Echocardiography (ECHO) - Postoperative reduction of left ventricular (LV) end-diastolic diameter of > 10 mm in an individual patient | in patients undergoing valve surgery 3-12 months after surgery
  in participants undergoing valve surgery within follow-up
Magnetic resonance imaging (MRI) - Postoperative improvement of left ventricular ejection fraction (LV EF) (all values) and/or reduction of left ventricular ejection fraction (LV EF) < 5% in an individual patient | in patients undergoing valve surgery 3-12 months after surgery
  in participants undergoing valve surgery within follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Radka Kockova, MD, PhD, Principal Investigator — Institute for Clinical and Experimental Medicine; Ales Linhart, Prof,MD,PhD, Study Director — General University Hospital; Hana Linkova, MD, PhD, Study Director — Faculty Hospital Kralovske Vinohrady; Martin Penicka, Study Director — VZW Cardiovascular Research Center Aalst
Locations (5):
- VZW Cardiovascular Research Center Aalst, Aalst, Belgium
- Czechia (4):
  - Karel Medilek, M.D., Hradec Králové
  - Institute for Clinical and Experimental Medicine, Prague
  - Faculty Hospital Kralovske Vinohrady, Prague
  - General University Hospital, Prague

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Iung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). [Guidelines on the management of valvular heart disease (version 2012). The Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)]. G Ital Cardiol (Rome). 2013 Mar;14(3):167-214. doi: 10.1714/1234.13659. No abstract available. Italian. PMID 23474606
- [Background] Aicher D, Fries R, Rodionycheva S, Schmidt K, Langer F, Schafers HJ. Aortic valve repair leads to a low incidence of valve-related complications. Eur J Cardiothorac Surg. 2010 Jan;37(1):127-32. doi: 10.1016/j.ejcts.2009.06.021. Epub 2009 Jul 29. PMID 19643618
- [Background] Smedsrud MK, Pettersen E, Gjesdal O, Svennevig JL, Andersen K, Ihlen H, Edvardsen T. Detection of left ventricular dysfunction by global longitudinal systolic strain in patients with chronic aortic regurgitation. J Am Soc Echocardiogr. 2011 Nov;24(11):1253-9. doi: 10.1016/j.echo.2011.08.003. Epub 2011 Sep 10. PMID 21908174
- [Background] Chaliki HP, Mohty D, Avierinos JF, Scott CG, Schaff HV, Tajik AJ, Enriquez-Sarano M. Outcomes after aortic valve replacement in patients with severe aortic regurgitation and markedly reduced left ventricular function. Circulation. 2002 Nov 19;106(21):2687-93. doi: 10.1161/01.cir.0000038498.59829.38. PMID 12438294
- [Background] Messroghli DR, Radjenovic A, Kozerke S, Higgins DM, Sivananthan MU, Ridgway JP. Modified Look-Locker inversion recovery (MOLLI) for high-resolution T1 mapping of the heart. Magn Reson Med. 2004 Jul;52(1):141-6. doi: 10.1002/mrm.20110. PMID 15236377
- [Background] Mewton N, Liu CY, Croisille P, Bluemke D, Lima JA. Assessment of myocardial fibrosis with cardiovascular magnetic resonance. J Am Coll Cardiol. 2011 Feb 22;57(8):891-903. doi: 10.1016/j.jacc.2010.11.013. PMID 21329834
- [Background] Reant P, Barbot L, Touche C, Dijos M, Arsac F, Pillois X, Landelle M, Roudaut R, Lafitte S. Evaluation of global left ventricular systolic function using three-dimensional echocardiography speckle-tracking strain parameters. J Am Soc Echocardiogr. 2012 Jan;25(1):68-79. doi: 10.1016/j.echo.2011.10.009. Epub 2011 Nov 13. PMID 22082980
- [Background] Russo C, Jin Z, Elkind MS, Rundek T, Homma S, Sacco RL, Di Tullio MR. Prevalence and prognostic value of subclinical left ventricular systolic dysfunction by global longitudinal strain in a community-based cohort. Eur J Heart Fail. 2014 Dec;16(12):1301-9. doi: 10.1002/ejhf.154. Epub 2014 Sep 11. PMID 25211239
- [Background] Kockova R, Kacer P, Pirk J, Maly J, Sukupova L, Sikula V, Kotrc M, Barciakova L, Honsova E, Maly M, Kautzner J, Sedmera D, Penicka M. Native T1 Relaxation Time and Extracellular Volume Fraction as Accurate Markers of Diffuse Myocardial Fibrosis in Heart Valve Disease - Comparison With Targeted Left Ventricular Myocardial Biopsy. Circ J. 2016 Apr 25;80(5):1202-9. doi: 10.1253/circj.CJ-15-1309. Epub 2016 Mar 17. PMID 26984717
- [Derived] Kockova R, Linkova H, Hlubocka Z, Medilek K, Tuna M, Vojacek J, Skalsky I, Cerny S, Maly J, Hlubocky J, Mizukami T, De Colle C, Penicka M. Multiparametric Strategy to Predict Early Disease Decompensation in Asymptomatic Severe Aortic Regurgitation. Circ Cardiovasc Imaging. 2022 Dec;15(12):e014901. doi: 10.1161/CIRCIMAGING.122.014901. Epub 2022 Dec 20. PMID 36538596
- See also: V1.4 MRmap software — http://sourceforge.net/projects/mrmap